CLINICAL TRIAL: NCT05342402
Title: Assessing the Feasibility of Somatosensory Rehabilitation and Pain Management Programs in Women With Provoked Vestibulodynia
Brief Title: Feasibility Study for Provoked Vestibulodynia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Principal Investigator, Mélanie Morin, Researcher and Full Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #2022-4357
Record Dates: First submitted 2022-04-16; First posted 2022-04-22 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Vestibulodynia
Keywords: Provoked Vestibulodynia; Pain; Allodynia; Somatosensory Rehabilitation
MeSH Terms: conditions — Vulvodynia; Pain; Hyperalgesia

STUDY DESIGN:
Intervention Model Description: Baseline evaluation - Randomization to Somatosensory Rehabilitation Program or Educational Pain Management Program (12 sessions within 12 weeks) - 2 weeks post-treatment evaluation - 3 months follow-up
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Somatosensory Rehabilitation Program (Experimental): Includes minimizing contact with the painful zone of the vulva and uses tactile stimulation at a tolerated distance from the vulva. Each participant will also receive advice on resuming sexual activities with vaginal penetration.
  Interventions: Other: Somatosensory Rehabilitation Program
- Educational Pain Management Program (PMP) (Active Comparator): Includes education on decreasing irritative contacts with the vulva and relaxation techniques. Each participant will also receive advice on resuming sexual activities with vaginal penetration.
  Interventions: Other: Educational Pain Management Program

INTERVENTIONS:
Other: Somatosensory Rehabilitation Program — Somatosensory rehabilitation program includes minimizing contact with the painful zone of the vulva and uses tactile stimulation at a tolerated distance from the vulva. Each participant will also receive advice on resuming sexual activities with vaginal penetration.
  Arms: Somatosensory Rehabilitation Program
Other: Educational Pain Management Program — Educational Pain Management Program includes education on decreasing irritative contacts with the vulva and relaxation techniques. Each participant will also receive advice on resuming sexual activities with vaginal penetration.
  Arms: Educational Pain Management Program (PMP)

SUMMARY:
The feasibility and acceptability of a somatosensory rehabilitation program and an educational pain management program will be investigated in women with provoked vestibulodynia. Forty-four women will be randomized into the two groups. The secondary objective is to explore the effects of the somatosensory rehabilitation program compared to the pain management program. Each participant will receive 12 weekly sessions with a physiotherapist.

The somatosensory rehabilitation program includes minimizing contact with the painful zone of the vulva and uses repeated tactile stimulation at a tolerated distance, proximal to the vulva. The pain management program includes teaching participants about vulvar hygiene, chronic pain mechanisms, relaxation techniques, and approaches to reduce skin irritations in painful regions. Participants in both groups will also receive advice on sexual function and steps toward resuming sexual activities with vaginal penetration.

Feasibility and acceptability outcomes will be assessed and analyzed using descriptive statistics for the adherence rates to treatment sessions and home exercises, the recruitment rate, retention rate, satisfaction, and adverse effects. The results will be compared to predetermined thresholds to determine the feasibility and acceptability of a future clinical trial.

Secondary measures will be assessed at baseline, two weeks after the treatment, and at three months follow-up. These outcomes will be assessed using validated questionnaires (pain, sexual function, global impression of change, psychological variables, quality of life) as well as evaluations of tactile and pressure sensitivity in vulvar regions using monofilaments, a 2-point aesthesiometer and an algometer. Linear mixed models for repeated measurements (2 groups, 3 measurement times) will be used to explore the treatment effects and will contribute to determining the feasibility of a future clinical trial.

Hypothesis and expected results: It is expected that both programs will meet the pre-determined criteria for acceptability and feasibility in women with provoked vestibulodynia. This study will provide guidance for a future randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of provoked vestibulodynia according to a standardized gynaecologic exam
2. Moderate to severe pain (≥5/10) located in the vulvar vestibule for at least 90% of vaginal penetrations or attempted vaginal penetrations or activities with pressure on the vagina for at least 3 months

Exclusion Criteria:

1. Other causes of vulvo-vaginal pain (e.g. spontaneous vulvovaginal pain not related to sexual intercourse/contact, dermatological condition, herpes, vulvo-vaginal atrophy)
2. Prior vulvo-vaginal surgery or radiotherapy
3. Post-menopausal status
4. Participant refusal to not use other treatments for the provoked vestibulodynia during the entire study (until 3 months post-treatment);
5. Other urogynecological condition (e.g. pelvic organs prolapse ≥3, current urinary/vaginal infection or in the last 3 months)
6. Prior use of Somatosensory Rehabilitation Program or Educational Pain Management Program
7. Current or past pregnancy in the last year;
8. Changes of medication that could influence pain perception (e.g. analgesic, antidepressant) in the last 3 months
9. Major psychological condition (e.g. depressive symptoms, anxiety) which can present a security issue for the participant
10. Other medical conditions that could interfere with the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Adherence rate to home exercises | From first to last session (baseline to 12th week)
  The adherence rate to home exercises for each treatment group will be assessed using a daily diary. The participants will record the frequency and duration of the exercises completed.
Patients' adherence rate to treatment sessions | From first to last session (baseline to 12th week)
  The patients' adherence to treatment sessions will be recorded in the participants' treatment files (present vs absent).
Adherence rate to assessment sessions | Baseline to 3 months post-treatment evaluation
  The adherence to assessment sessions (present vs absent) will be recorded in the participants' assessment files. The reasons for absences will be documented.
Retention rate | Baseline to 3 months post-treatment evaluation
  The retention rate will be assessed by calculating the ratio of participants who stay in the study until the post-intervention and 3-month follow-up assessments. Reasons for dropouts will be collected.
Recruitment rate | At baseline only (during the recruitement period)
  The recruitment rate will be recorded as the average number of participants recruited per month as well as the participant accrual rate (participants enrolled / participants screened for diagnosis). Reasons for refusing to participate will be documented if the participant consents to inform the study's research team.
Therapists treatment adherence | From first to last session (baseline to 12th week)
  The therapists' treatment adherence will be assessed within the therapists' files to verify that all the interventions' key components were applied and respected.

SECONDARY OUTCOMES:
Intervention Acceptability Questionnaire | At 2-week post-treatment and at 3 months post-treatment
  The Intervention Acceptability Questionnaire explores the participants' acceptability of the interventions. This questionnaire consists of 4 items measured on a VAS scale (Minimum value: 0; Maximum Value: 10). Each item is analyzed separately, with a greater score meaning higher acceptability of the intervention. This outcome measure will contribute to identifying factors limiting the acceptability of each program.
Credibility and Expectancy Questionnaire | At baseline only (before the initiation of the treatment)
  The Credibility and Acceptability Questionnaire explores the credibility and the participants' expectancy for the interventions. This questionnaire consists of 3 items: two items are measured on a 9-point Likert scale (Minimum value: 1; Maximum Value: 9) and one item is measured in percentages (Minimum: 0, Maximum: 100%). Each item is analyzed separately, with a greater score meaning higher credibility.
Patients' Global Impression of Change and Satisfaction | At 2-week post-treatment and 3 months post-treatment
  These two items will determine patient self-reported improvement and satisfaction regarding the effects of the intervention on pain (Patient's Global Impression of Change and Satisfaction). The Patient's Global Impression of Change contains two items that address change in pain and quality of sexual life. It is assessed on a 7-point scale ranging from "very much worse" to "very much improvement". The Satisfaction will be assessed with a single item on an 11-point Likert scale (Minimum: 0, Maximum: 10). A greater score means higher satisfaction. This outcome measure explores the acceptability of the interventions by assessing the extent to which the intervention is perceived as likely to achieve its purpose.
Self-Efficacy Question | At baseline, 6 week after the initiation of treatment, and at the last treatment (12th week)
  A single item included in the participant's diary will assess at which point the participant feels she is confident and self-sufficient in being able to apply the exercises and advice. This item is measured on a VAS scale (Minimum: 0, Maximum: 10) with a greater score meaning higher confidence in being self-sufficient in applying the exercises and advice. This outcome measure will explore self-efficacy regarding the interventions.
Adverse events | 2-week and 3 months post-treatment
  The adverse events will be noted in the participant's daily diary and in the treatment files.
Pain intensity during intercourse (Numerical Rating Scale) | Changes from pre- to 2-week post-treatment, from 2-week post-treatment to 3-month post-treatment, and from pre-treatment to 3-month post-treatment
  Pain during intercourse will be assessed using a numeric rating scale (NRS) ranging from 0 to 10, where 0 is no pain at all, and 10 is the worst pain ever.
Pain quality (McGill-Melzack questionnaire-short form) | Change in the scores from pre- to 2-week post-treatment, from 2-week post-treatment to 3-month post-treatment, and from pre-treatment to 3-month post-treatment
  The McGill-Melzack questionnaire- short form consists of 15 items that assess the sensory, affective and evaluative components of pain. Items are scored on a 4-point scale with the endpoints (0) no pain at all and (3) severe pain. Minimum value: 0, Maximum value: 45, with more elevated scores meaning higher pain.
Vulvar sensitivity | Change in the scores from pre- to 2-week post-treatment, from 2-week post-treatment to 3-month post-treatment, and from pre-treatment to 3-month post-treatment
  Gradual pressure (1 to 1000 g) will be applied to three distinct points of the vestibule at the 3, 6 and 9 o'clock positions. Each of these pressure points will be applied randomly (e.g. 3,6,9 or 3,9,6 or 6,9,3.). During this procedure, each participant will be asked to indicate when they start to feel pain (pain threshold) and subsequently the maximal pressure that can be tolerated (pain tolerance). A higher result means a more elevated pain threshold and a higher pain tolerance.
Vulvar tactile allodynia area | Change in the surface from pre- to 2-week post-treatment, from 2-week post-treatment to 3-month post-treatment, and from pre-treatment to 3-month post-treatment
  A force of 15g will be applied using a monofilament in the vulvar region in order to outline the borders of the allodynia (hypersensitivity to tactile stimuli) surface. The width and length of the surface will be measured with a graduated cotton swab (ruler). The surface will be computed by multiplying its width by its length (squared centimeters). This method of assessing allodynia severity is described within the Somatosensory Rehabilitation Method Handbook. A higher value indicates a greater area with tactile allodynia.
Vulvar tactile alllodynia severity | Change in the surface from pre- to 2-week post-treatment, from 2-week post-treatment to 3-month post-treatment, and from pre-treatment to 3-month post-treatment
  A series of seven monofilaments (0.02g, 0.4g, 0.7g, 1.5g, 4.0g, 8.0g, 15.0g) will be applied to the outside border of the vulvar vestibule to find the smallest force that causes an increase in pain. This method of assessing allodynia severity is described within the Somatosensory Rehabilitation Method Handbook. A lower result indicates more severe allodynia.
Vulvar tactile sensibility | Change in the surface from pre- to 2-week post-treatment, from 2-week post-treatment to 3-month post-treatment, and from pre-treatment to 3-month post-treatment
  Once the allodynia has resolved, the smallest perceived force will be measured by applying monofilaments in a decreasing order (force) to the outside border of the vulvar vestibule (Max: 29g; Min: 0.005g). A lower force value indicates better tactile sensibility.
Two-point discrimination test | Change in the surface from pre- to 2-week post-treatment, from 2-week post-treatment to 3-month post-treatment, and from pre-treatment to 3-month post-treatment
  The two-point discrimination test assesses an integrative aspect of tactile sensibility. Once the allodynia has resolved, a 2-point stainless steel aesthesiometer will be applied with one point on the vulvar vestibule border and the other point outside this area. It will be applied at variable and decreasing distances. The result is the smallest distance between the two points at which the person can discriminate if one or two points are being applied (Minimum: 1mm, Maximum: 100mm). A smaller value suggests tactile perception of a higher quality.
Female Sexual Function Index (FSFI) | Change in the scores from pre- to 2-week post-treatment, from 2-week post-treatment to 3-month post-treatment, and from pre-treatment to 3-month post-treatment
  The Female Sexual Function Index (FSFI) is a multidimensional measure of sexual function evaluating desire, arousal, lubrication, orgasm, satisfaction and pain. This 19-item questionnaire explores changes in sexual function with a Likert scale ranging from 0 (or 1) to 5. The overall score has a minimum value of 2 and a maximum value of 36. Lower scores mean worse outcomes (low sexual function).
Female Sexual Distress Scale (FSDS) | Change in the scores from pre- to 2-week post-treatment, from 2-week post-treatment to 3-month post-treatment, and from pre-treatment to 3-month post-treatment
  The FSDS 13-item questionnaire explores sexually related personal distress in women. Each item is assessed on a 5-point Likert scale from 0 (never) to 5 (always). The total score ranges from a minimum value of 0 to a maximum value of 100. Higher scores mean worse outcomes (greater sexually related distress).
Pain Anxiety Symptoms Scale (PASS-20) | Change in the scores from pre- to 2-week post-treatment, from 2-week post-treatment to 3-month post-treatment, and from pre-treatment to 3-month post-treatment
  The PASS-20 is a 20-item questionnaire that explores fear and anxiety responses specific to pain. Each item is assessed on a 6-point Likert scale from 0 (never) to 4 (always). The total score ranges from a minimum value of 0 to a maximum value of 52. Higher scores mean worse outcomes (greater fear of pain).
Pain Catastrophizing Scale (PCS) | Change in the scores from pre- to 2-week post-treatment, from 2-week post-treatment to 3-month post-treatment, and from pre-treatment to 3-month post-treatment
  Pain catastrophizing will be assessed using the PCS, which consists of 13 items measuring exaggerated negative thoughts and feelings about the meaning of pain. Items are scored on a 5-point scale with the endpoints (0) not at all and (4) all the time. Minimum value: 0, Maximum value: 52, higher scores mean worse outcomes (greater pain catastrophizing).
Beck Depression Inventory questionnaire (BDI-II) | Change in the scores from pre- to 2-week post-treatment, from 2-week post-treatment to 3-month post-treatment, and from pre-treatment to 3-month post-treatment
  Depression or depression symptoms will be measured with the Beck Depression Inventory-II (BDI-II). The BDI-II is comprised of 21 items, with scores for most items ranging from 0 (low intensity) to 3 (high intensity). The maximum total score is 63. Scores above 10 meet the threshold for depression. Higher scores mean more severe depression.
Vaginal Penetration Cognition Questionnaire (VPCQ) | Change in the scores from pre- to 2-week post-treatment, and from pre-treatment to 3-month post-treatment
  The VPCQ is a 40-item questionnaire that assesses cognitions regarding vaginal penetration in women. Items are scored on a 6-point scale with the end points (0) never and (6) always. Five aspects of vaginal penetration cognition are assessed: control cognitions, catastrophic and pain cognitions, self-image cognitions, positive cognitions, and genital incompatibility cognitions. Higher scores show higher levels of perceived penetration control.
12-item Short Form Survey (SF-12 v2) | Change in the scores from pre- to 2-week post-treatment, from 2-week post-treatment to 3-month post-treatment, and from pre-treatment to 3-month post-treatment
  The SF-12 questionnaire assesses the impact of health on an individual's everyday life and quality of life. The second version of the SF-12 will be used. Scores range from 0 (minimum) to 100 (maximum). Higher scores indicate better physical and mental health.

OTHER OUTCOMES:
Short-Leeds Assessment for Neuropathic Symptoms and Signs (S-LANSS) | At baseline only (before the initiation of the treatment)
  The S-LANSS 7-item questionnaire assesses the presence of neuropathic symptoms and signs. The dichotomous answers have different weights in the total score with the absence of the sign/symptom valued at 0 and the presence of the sign/symptom valued between 1 and 5 points. Scores range from 0 (minimum) to 24 (maximum). Scores of 12 or greater suggest pain of a predominantly neuropathic origin. The proportion of neuropathic symptoms and signs in each group will be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

REFERENCES:
- See also: Facebook page — https://www.facebook.com/pages/Laboratoire-de-recherche-en-urogyn%C3%A9cologie/277240805641504?fref=ts
- See also: Laboratory Web page — http://www.lab-urogyn.com/